CLINICAL TRIAL: NCT03517254
Title: Effect of Oral Complementation of Glutamine on Knee Strengths Indicators in Adult Patients With Anterior Cruciate Ligament Reconstruction. A Double-blinded, Randomized Controlled Trial
Brief Title: Use of Glutamine for Recovery Muscle Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Sandra Hernández Valencia, Principal investigator, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 47/16
Record Dates: First submitted 2018-04-05; First posted 2018-05-07 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Glutamine,
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glutamine and strength training program (Experimental): Three times per week, standardized and supervised resistance training by physicians will be conducted at the National Institute of Rehabilitation for 6 weeks of follow up. At the beginning and at the end of the training session, the experimental group will receive by mouth 10 grams of glutamine dissolved in 120 milliliters of water, all participants and team of researchers will not be aware of the supplement.
  Interventions: Dietary Supplement: Glutamine; Other: Strength training program; Other: Dietary recommendations
- Placebo and strength training program (Placebo Comparator): Three times per week a standardized and supervised resistance training by physicians will be conducted at the National Institute of Rehabilitation for 6 weeks after discharge. At the beginning and at the end of the training session, the placebo group will receive by mouth10 grams of maltodextrin dissolved in 120 milliliters of water. All participants and team of researchers will not be aware of the supplement content.
  Interventions: Other: Strength training program; Other: Placebo; Other: Dietary recommendations

INTERVENTIONS:
Dietary Supplement: Glutamine — At the beginning and at the end of the training session, the experimental group will receive by mouth 15 grams of glutamine dissolved in 120 milliliters of water. The aminoacid will be inside gray envelopes.
  Other Names: Glutapak 10
  Arms: Glutamine and strength training program
Other: Strength training program — One training session consists of 20 minutes of warm-up, 40 to 60 minutes of aerobic and anaerobic exercises and 15 minutes of cooling down. The exercises of the lower part of the body consist in 3 sets of 10 repetitions for healthy knee, and 12 repetitions for knee with anterior cruciate ligament reconstruction in a modular leg press, leg curl and leg extension machine.
Other: Placebo — Maltodextrin powder to mimic glutamine,
  Arms: Placebo and strength training program
Other: Dietary recommendations — All participants, irrespective of the supplement that they receive, will be closely monitored by a nutritionist, who will give dietary recommendations to standardize protein consumption (1.2 gr/kg weight). Status nutritional will be assessed according to BMI ( 19.9-24.9, 25-29.9).

SUMMARY:
After an Anterior Cruciate Ligament Reconstruction by surgery, the most important muscle of the knee, called quadriceps femoral, loses strength in more than 60% of cases, which if not corrected can progress to osteoarthritis in up to 80% of patients, compromising their quality of life.

The main treatment for loss of muscle strength in these patients is rehabilitation which includes strength and endurance exercises.However, in some cases, amino acids such as Glutamine (Gln) have been employed as an aid to recover muscle strength, but the evidence on this topic is not consistent and is inconclusive. Therefore, the main purpose of this study is to investigate if the oral complementation with Glutamine in combination with strength and resistance training can improve the muscle strength of the quadriceps femoral in patients with anterior cruciate ligament reconstruction compared with those receiving a placebo after six weeks of intervention.

DETAILED DESCRIPTION:
The study design is a randomized, double-blind and controlled trial. A total of 50 adult men will be recruited from medical departments of the National Institute of Rehabilitation in Mexico City.

Patients: Fifty men 20 to 50 years old, between 15 to 19 weeks after surgical reconstruction of anterior cruciate ligament and moderate loss of muscle strength of knee (assessment with computerized dynamometer), will be recruited from the Sport Rehabilitation department, and the treatment will be carried out in the Sport Medicine area, both of the National Institute of Rehabilitation in Mexico City. Patients with diabetes, obesity, hypertension, kidney or liver diseases or with glucocorticoid treatment, and athletes will not be included.

Intervention: The sample will be randomized in two groups. At the beginning and at the end of the training session, the experimental group will receive 10 grams of glutamine, and the control group will receive 10 grams of placebo (maltodextrin), both dissolved in 120 milliliters of water and all participants will not be aware of the supplement content.

Both groups will participate in the same standardized resistance training program, to ensure progression (or regression if necessary) to all training components and adherence to the intervention, each participant will do the training program in a therapeutic gym of Sport Medicine area three times per week, during 6 weeks of follow-up. One training session consists of 20 minutes of warm-up, 40 to 60 minutes of aerobic and anaerobic exercises and 15 minutes of cooling down. The exercises of the lower part of the body consist in 3 sets of 10 repetitions for healthy knees, and 12 repetitions for knees with anterior cruciate ligament reconstruction in a modular leg press, leg curl and leg extension machine.

All participants, irrespective of the supplement that they receive, will be closely monitored by a physician specialist in Sport Medicine and a nutritionist, who will give a dietary program to standardize protein consumption. Status nutritional will be assessed according to Body Mass Index [(BMI) 19.9-24.9, 25-29.9].

Muscle strength will be measured by a computer dynamometer. The reliability of the dynamometry will be evaluated by Intraclass Correlation Coefficient (ICC). Thigh circumference will be measured by a anthropometric technique (Nutritionists certified by the International Society for the Advance of Kinanthropometry in level one, will carry out the measurement). Fasting glucose, lipid profile and liver function test will be carried out in the clinical laboratory of National Institute of Rehabilitation. The measurements are going to be held twice; before the first training session, and 6 weeks after.

For each participant the study duration will start in the first training session until 6 weeks after. Endpoints assessments will be performed at baseline (2 days before starting the training program) and after 6 weeks of follow-up (2 days after the last training session). Data will be collected by study investigators blinded to the allocation of the participants.

Comparison: The control group will receive maltodextrin powder (placebo) dissolved in 120 milliliters of water. The placebo will be inside gray envelopes, in the same manner that the glutamine was administered.

Outcomes: The main outcome is to change the strength of quadriceps femoris (assessment by isokinetic dynamometer).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 15 to 19 weeks after surgical reconstruction of anterior cruciate ligament
* Moderate loss of muscle strength of knee (assessment with computerized dynamometer)
* Perform the training sessions in the hospital
* No athletes
* Index Body Mass: 20 - 30 kg/m²
* Without consumption of supplements based on amino acids in the last 6 months
* To sign informed consent letter

Exclusion Criteria:

* Diabetes mellitus I or 2
* Liver and renal diseases
* Dyslipidemia
* Glucocorticoid consumption
* Active cancer
* Glutamine allergy or intolerance
* Planning to lose weight/go on special diet

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in torque peak of quadriceps femoris and hamstring | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up (1 day after the last training session)
  Measurement by computer dynamometer and expressed in Newton/meters at 60° angular speed.
Change hamstring/quadriceps ratio | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up (1 day after the last training session)
  Measurement by computer dynamometer and expressed in percentages at 60° angular speed.

SECONDARY OUTCOMES:
Change in thigh circumference (In operated knee and the non-operated knee) | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up (1 day after the last training session)
  Thigh circumference (centimeters) evaluated by fiberglass tape measure according to the technique that has been established by the International Society for the Advancement of Kinanthropomethry (ISAK).
Energy intake | Baseline (admission to Sport Medicine), 3 and 6 weeks after the follow-up]
  Dietary interviews twice (24-h recall interviews) (Energy Kcal)
Protein intake | Baseline (admission to Sport Medicine), 3 and 6 weeks after the follow-up]
  Dietary interviews twice (24-h recall interviews) (protein, g/kg)
Changes in blood glucose levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 8 hours of fasting. The quantification of blood glucose levels will be through the hexokinase method, which is used by Dimension clinical chemistry system.
Changes in total blood cholesterol levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting. The quantification of total blood cholesterol levels will be through the CHOL method, which is used by Dimension clinical chemistry system.
Changes in blood High Density Lipoprotein-Cholesterol (HDL-C) levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting. The quantification of blood HDL-C levels will be through AHDL-Method, which is used by Dimension clinical chemistry system.
Changes in blood Low density Lipoprotein-Cholesterol (LDL-C) levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting. The quantification of blood LDL-C levels will be through ALDL-Method, used by Dimension clinical chemistry system.
Changes in blood triglycerides levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting. The quantification of blood triglycerides levels will be through TGL-Method, used by Dimension clinical chemistry system.
Changes in blood Aspartate aminotransferase (AST) levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting. The quantification of blood Aspartate aminotransferase (AST) levels will be through AST-Method, used by Dimension clinical chemistry system.
Changes in blood alanine aminotransferase (ALT) levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting. The quantification of blood Alanine aminotransferase (ALT) levels will be through ALTI-Method, used by Dimension clinical chemistry system.
Changes in blood Alkaline phosphatase (ALP) levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting, for the quantification of blood Alkaline phosphatase (ALP) levels through method used by Dimension clinical chemistry system.
Changes in blood Gamma-glutamyl transferase (GGT) levels | Baseline (admission to Sport Medicine) and 6 weeks after the follow-up
  A sample of 5 milliliters of blood will be taken from patients with 12 hours of fasting. The quantification of blood Gamma-glutamyl transferase (GGT) levels will be through GGT-Method, used by Dimension clinical chemistry system.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Moreno Altamirano, PhD, Study Director — Universidad Nacional Autonoma de Mexico
Locations (1):
- Instituto Nacional de Rehabilitación, Mexico City, Mexico

REFERENCES:
- [Background] Nordenvall R, Bahmanyar S, Adami J, Mattila VM, Fellander-Tsai L. Cruciate ligament reconstruction and risk of knee osteoarthritis: the association between cruciate ligament injury and post-traumatic osteoarthritis. a population based nationwide study in Sweden, 1987-2009. PLoS One. 2014 Aug 22;9(8):e104681. doi: 10.1371/journal.pone.0104681. eCollection 2014. PMID 25148530
- [Background] Frobell RB, Roos EM, Roos HP, Ranstam J, Lohmander LS. A randomized trial of treatment for acute anterior cruciate ligament tears. N Engl J Med. 2010 Jul 22;363(4):331-42. doi: 10.1056/NEJMoa0907797. PMID 20660401
- [Background] Adams D, Logerstedt DS, Hunter-Giordano A, Axe MJ, Snyder-Mackler L. Current concepts for anterior cruciate ligament reconstruction: a criterion-based rehabilitation progression. J Orthop Sports Phys Ther. 2012 Jul;42(7):601-14. doi: 10.2519/jospt.2012.3871. Epub 2012 Mar 8. PMID 22402434
- [Background] Hsiao SF, Chou PH, Hsu HC, Lue YJ. Changes of muscle mechanics associated with anterior cruciate ligament deficiency and reconstruction. J Strength Cond Res. 2014 Feb;28(2):390-400. doi: 10.1519/JSC.0b013e3182986cc1. PMID 23669818
- [Background] Thomas AC, Villwock M, Wojtys EM, Palmieri-Smith RM. Lower extremity muscle strength after anterior cruciate ligament injury and reconstruction. J Athl Train. 2013 Sep-Oct;48(5):610-20. doi: 10.4085/1062-6050-48.3.23. Epub 2013 Apr 18. PMID 24067150
- [Background] Zuka-Nowak K, Ogrodzka K, Chwala W, Niedzwiedzki L, Niedzwiedzki T. Kinetic and kinematic characteristics of natural velocity gait in anterior cruciate ligament-deficient patients. Int J Rehabil Res. 2013 Jun;36(2):152-61. doi: 10.1097/MRR.0b013e32835c79c5. PMID 23238669
- [Background] Orri JC, Darden GF. Technical report: Reliability and validity of the iSAM 9000 isokinetic dynamometer. J Strength Cond Res. 2008 Jan;22(1):310-7. doi: 10.1519/JSC.0b013e31815fa2c8. PMID 18296991
- [Background] Risberg MA, Lewek M, Snyder-MacKler L. A systematic review of evidence for anterior cruciate ligament rehabilitation: how much and what type?. Phys Ther Sport (5): 125-145, 2004
- [Background] Trees AH, Howe TE, Dixon J, White L. Exercise for treating isolated anterior cruciate ligament injuries in adults. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD005316. doi: 10.1002/14651858.CD005316.pub2. PMID 16235401
- [Background] Eitzen I, Moksnes H, Snyder-Mackler L, Risberg MA. A progressive 5-week exercise therapy program leads to significant improvement in knee function early after anterior cruciate ligament injury. J Orthop Sports Phys Ther. 2010 Nov;40(11):705-21. doi: 10.2519/jospt.2010.3345. PMID 20710097
- [Background] Cermak NM, Res PT, de Groot LC, Saris WH, van Loon LJ. Protein supplementation augments the adaptive response of skeletal muscle to resistance-type exercise training: a meta-analysis. Am J Clin Nutr. 2012 Dec;96(6):1454-64. doi: 10.3945/ajcn.112.037556. Epub 2012 Nov 7. PMID 23134885
- [Background] Pasiakos SM, McLellan TM, Lieberman HR. The effects of protein supplements on muscle mass, strength, and aerobic and anaerobic power in healthy adults: a systematic review. Sports Med. 2015 Jan;45(1):111-31. doi: 10.1007/s40279-014-0242-2. PMID 25169440
- [Background] Holm L, Esmarck B, Mizuno M, Hansen H, Suetta C, Holmich P, Krogsgaard M, Kjaer M. The effect of protein and carbohydrate supplementation on strength training outcome of rehabilitation in ACL patients. J Orthop Res. 2006 Nov;24(11):2114-23. doi: 10.1002/jor.20147. PMID 16917926
- [Background] Eichner ER. Glutamine supplementation: overstaying its welcome. Curr Sports Med Rep. 2013 Jul-Aug;12(4):211-2. doi: 10.1249/JSR.0b013e31829b54c8. No abstract available. PMID 23851404
- [Background] Mason BC, Lavallee ME. Emerging supplements in sports. Sports Health. 2012 Mar;4(2):142-6. doi: 10.1177/1941738111428127. PMID 23016081
- [Background] Agostini F, Biolo G. Effect of physical activity on glutamine metabolism. Curr Opin Clin Nutr Metab Care. 2010 Jan;13(1):58-64. doi: 10.1097/MCO.0b013e328332f946. PMID 19841583
- [Background] Piattoly T, Parish TR, Welsch MA. L-Glutamine Supplementation: effects on endurance, power and recovery. Curr Top Nutraceutical Res 11(1-2): 55-62, 2013.
- [Background] Hernandez Valencia SE, Mendez Sanchez L, Clark P, Moreno Altamirano L, Mejia Arangure JM. [GLUTAMINE AS AN AID IN THE RECOVERY OF MUSCLE STRENGTH: SYSTEMATIC REVIEW OF LITERATURE]. Nutr Hosp. 2015 Oct 1;32(4):1443-53. doi: 10.3305/nh.2015.32.4.9321. Spanish. PMID 26545503
- [Background] Legault Z, Bagnall N, Kimmerly DS. The Influence of Oral L-Glutamine Supplementation on Muscle Strength Recovery and Soreness Following Unilateral Knee Extension Eccentric Exercise. Int J Sport Nutr Exerc Metab. 2015 Oct;25(5):417-26. doi: 10.1123/ijsnem.2014-0209. Epub 2015 Mar 26. PMID 25811544
- [Background] Waddell D Fredricks K. Effects of a Glutamine Supplement on the Skeletal Muscle Contractile Force of Mice. Am J Undergraduate Res 4:11-18, 2005.